CLINICAL TRIAL: NCT02397122
Title: The Adjunctive Effect of Platelet Rich Fibrin to Connective Tissue Graft in the Treatment of Buccal Recession Defects. Results of a Randomized Parallel Group Controlled Trial
Brief Title: Platelet-rich Fibrin and Connective Tissue Graft in Recession Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, H. Gencay Keceli, DDS, PhD, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KirikkaleU
Record Dates: First submitted 2015-02-13; First posted 2015-03-24 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRF+CAF+CTG (Experimental): platelet-rich fibrin + coronally advanced flap + connective tissue graft
  Interventions: Biological: platelet-rich fibrin; Procedure: connective tissue graft; Procedure: coronally advanced flap
- CAF+CTG (Active Comparator): coronally advanced flap + connective tissue graft
  Interventions: Procedure: connective tissue graft; Procedure: coronally advanced flap

INTERVENTIONS:
Biological: platelet-rich fibrin — autologous platelet-rich fibrin was isolated from venous blood of each patient by defined centrifugation methods
  Arms: PRF+CAF+CTG
Procedure: connective tissue graft — connective tissue graft was harvested from the palatal region of each patient by single incision method
Procedure: coronally advanced flap — buccal gingival flap was raised by sharp-blunt-sharp dissection and positioned coronally to cover connective tissue graft (and platelet-rich fibrin gel)

SUMMARY:
The aim of the trial is to evaluate the effectiveness of coronally advanced flap (CAF)+connective tissue graft(CTG)+platelet-rich fibrin(PRF) combination in Miller I and II recession treatment by comparing with CAF+CTG. 40 patients were surgically treated either with CAF+CTG+PRF (test group) or CAF+CTG (control group). Clinical parameters of plaque index (PI), gingival index (GI), vertical recession (VR), probing depth (PD), attachment level (AL), keratinized tissue width (KTW), horizontal recession (HR), MGJ localization (L-MGJ), tissue thickness (TT) were recorded at baseline, 3 months (PS1) and 6 months (PS2) post-surgery. Root coverage (RC), complete RC (CRC), attachment gain (AG), and keratinized tissue change (KTC) were also calculated.

DETAILED DESCRIPTION:
Given the encouraging effects of platelet-rich fibrin (PRF) in healing and regeneration, it has been hypothesized that PRF might develop the outcomes obtained with coronally advanced flap (CAF)+connective tissue graft(CTG). Therefore, it was aimed to evaluate the effectiveness of CAF + CTG + PRF in Miller Class I and II recession defect treatment by comparing the outcomes with CAF + CTG in a preliminary, controlled, randomized clinical trial (RCT) with a 6-month follow-up. The study was conducted with 40 patients randomly grouped in half shares into indicated study groups. After phase I therapy, clinical variables including plaque index (PI), gingival index (GI), vertical recession (VR), probing depth (PD), attachment level (AL), keratinized tissue width (KTW), horizontal recession (HR), MGJ localization (L-MGJ), tissue thickness (TT) were recorded. The surgical sites were prepared by using sulcular and adjacent vertical incisions and CTGs were harvested from the palatal regions. Different from CAF+CTG group, PRF was prepared by obtaining 10 ml venous blood, centrifugation and extraction of the gel containing highly concentrated platelet cells in CAF+CTG+PRF patients. Then the gel was placed over the exposed root surface in the same group. The CAF was primarily closed and postoperative instructions were given. After suture removal at second postoperative week, the patients were followed-up by monthly recall visits. Same periodontal clinical variables were recorded 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Single Miller type I or II recession defect ≥ 3 mm localized to anterior/premolar area
* No alveolar bone loss
* Identifiable cemento-enamel junction
* Probing depth ≤3mm

Exclusion Criteria:

* Smoking
* Pregnancy
* History of periodontal surgery in last two years
* Mobility
* Excessive occlusal contacts
* Caries
* Loss of vitality

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-eight patients that did not comply with the inclusion criteria were not chosen for the study
Groups:
- CAF+CTG+PRF: platelet-rich fibrin + coronally advanced flap + connective tissue graft
  platelet-rich fibrin: autologous platelet-rich fibrin was isolated from venous blood of each patient by defined centrifugation methods
  connective tissue graft: connective tissue graft was harvested from the palatal region of each patient by single incision method
  coronally advanced flap: buccal gingival flap was raised by sharp-blunt-sharp dissection and positioned coronally to cover connective tissue graft (and platelet-rich fibrin gel)
- CAF+CTG: coronally advanced flap + connective tissue graft
  connective tissue graft: connective tissue graft was harvested from the palatal region of each patient by single incision method
  coronally advanced flap: buccal gingival flap was raised by sharp-blunt-sharp dissection and positioned coronally to cover connective tissue graft
Period: Overall Study
Arm/Group | CAF+CTG+PRF | CAF+CTG
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CAF+CTG+PRF: A computer-generated randomization scheme (simple randomization without any blocking) was used to assign 20 patients into each study groups with an allocation ratio of 1:1 The surgical sites were prepared by using sulcular and adjacent vertical incisions and CTGs were harvested from the palatal regions. Different from CAF+CTG group, PRF was prepared by obtaining 10 ml venous blood, centrifugation and extraction of the gel containing highly concentrated platelet cells in CAF+CTG+PRF patients. Then the gel was placed over the exposed root surface in the same group and the CAF was primarily closed.
- CAF+CTG: A computer-generated randomization scheme (simple randomization without any blocking) was used to assign 20 patients into each study groups with an allocation ratio of 1:1 The surgical sites were prepared by using sulcular and adjacent vertical incisions and CTGs were harvested from the palatal regions. CTG was placed over the exposed root surface and the CAF was primarily closed onto it.
- Total: Total of all reporting groups
Arm/Group | CAF+CTG+PRF | CAF+CTG | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.80 (7.85) | 39.65 (6.46) | 40.72 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 8 | 5 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Vertical Recession
Description: Measured from cementoenamel junction to margin of the gingiva by periodontal probe
Time Frame: Baseline, 6 weeks and 6 months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- CAF+CTG: platelet-rich fibrin + coronally advanced flap + connective tissue graft
  platelet-rich fibrin: autologous platelet-rich fibrin was isolated from venous blood of each patient by defined centrifugation methods
  connective tissue graft: connective tissue graft was harvested from the palatal region of each patient by single incision method
  coronally advanced flap: buccal gingival flap was raised by sharp-blunt-sharp dissection and positioned coronally to cover connective tissue graft (and platelet-rich fibrin gel)
Arm/Group | PRF+CAF+CTG | CAF+CTG
Number analyzed (Participants) | 20 | 20
mm
  Baseline | 3.35 (0.43) | 3.20 (0.34)
  6 weeks | 0.38 (0.54) | 0.65 (0.59)
  6 months | 0.35 (0.52) | 0.65 (0.59)
Statistical Analysis 1: Comparison: PRF+CAF+CTG vs CAF+CTG; Baseline; Test type: Superiority; p = 0.259, Mann-Whitney
Statistical Analysis 2: Comparison: PRF+CAF+CTG vs CAF+CTG; 6 weeks; Test type: Superiority; p = 0.097, Mann-Whitney
Statistical Analysis 3: Comparison: PRF+CAF+CTG vs CAF+CTG; 6 months; Test type: Superiority; p = 0.070, Mann-Whitney U — <0.05

2. Secondary Outcome: Horizontal Recession
Description: measured horizontally between two borders of the recession at the line tangential to cementoenamel junction by periodontal probe
Time Frame: Baseline, 6 weeks and 6 months
Population: Data pertaining to 20 patients from each group were analysed after completing 6 months period
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- CAF+CTG: platelet-rich fibrin + coronally advanced flap + connective tissue graft
  platelet-rich fibrin: autologous platelet-rich fibrin was isolated from venous blood of each patient by defined centrifugation methods
  connective tissue graft: connective tissue graft was harvested from the palatal region of each patient by single incision method
  coronally advanced flap: buccal gingival flap was raised by sharp-blunt-sharp dissection and positioned coronally to cover connective tissue graft
Arm/Group | CAF+CTG+PRF | CAF+CTG
Number analyzed (Participants) | 20 | 20
mm
  Baseline | 3.8 [2 to 5] | 3 [2 to 5]
  6 weeks | 0 [0 to 3] | 1 [0 to 3]
  6 months | 0 [0 to 3] | 1 [0 to 2]
Statistical Analysis 1: Comparison: CAF+CTG+PRF vs CAF+CTG; Baseline; Test type: Superiority; p = 0.067, Mann-Whitney
Statistical Analysis 2: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 weeks; Test type: Superiority; p = 0.130, Mann-Whitney
Statistical Analysis 3: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 months; Test type: Superiority; p = 0.128, Mann-Whitney U — <0.05

3. Secondary Outcome: Probing Depth
Description: measured from margin of the gingiva to gingival sulcus base by periodontal probe
Time Frame: Baseline, 6 weeks and 6 months
Population: Data pertaining to 20 patients from each group were analysed after completing 6 months period
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- CAF+CTG+PRF: A computer-generated randomization scheme (simple randomization without any blocking) was used to assign 20 patients into each study groups with an allocation ratio of 1:1. After phase I therapy, the patients were surgically treated with coronally advanced flap (CAF)+connective tissue graft(CTG)+platelet-rich fibrin(PRF). Surgical incisions involving sulcular and adjacent vertical incisions were made and split-full-split flaps were elevated. PRF was prepared from 10 ml venous blood and the gel part was placed under CTG harvested from the palate. Flap was coronally advanced and CTG+PRF was completely closed. Extraoral cold compress and analgesic plus antiinflammatory drugs (Ibuprofen, 100 mg, twice a day) were given for pain and edema control. Toothbrushing in the surgical region was prohibited for 4 weeks; instead, antiseptic solution (Chlorhexidine gluconate) was prescribed.
- CAF+CTG: A computer-generated randomization scheme (simple randomization without any blocking) was used to assign 20 patients into each study groups with an allocation ratio of 1:1. After phase I therapy, the patients were surgically treated with coronally advanced flap (CAF)+connective tissue graft(CTG). Surgical incisions involving sulcular and adjacent vertical incisions were made and split-full-split flaps were elevated. CTG was harvested from the palate and placed over the recession defect. Flap was coronally advanced and CTG was completely closed. Extraoral cold compress and analgesic plus antiinflammatory drugs (Ibuprofen, 100 mg, twice a day) were given for pain and edema control. Toothbrushing in the surgical region was prohibited for 4 weeks; instead, antiseptic solution (Chlorhexidine gluconate) was prescribed.
Arm/Group | CAF+CTG+PRF | CAF+CTG
Number analyzed (Participants) | 20 | 20
mm
  Baseline | 1 [1 to 2] | 1 [1 to 2]
  6 weeks | 1 [1 to 1] | 1 [1 to 2]
  6 months | 1 [1 to 1] | 1 [1 to 2]
Statistical Analysis 1: Comparison: CAF+CTG+PRF vs CAF+CTG; Baseline; Test type: Superiority; p = 0.298, Mann-Whitney
Statistical Analysis 2: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 weeks; Test type: Superiority; p = 0.152, Mann-Whitney
Statistical Analysis 3: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 months; Test type: Superiority; p = 0.317, Mann-Whitney U — <0.05

4. Secondary Outcome: Attachment Level
Description: measured from cementoenamel junction to gingival sulcus base by periodontal probe
Time Frame: Baseline, 6 weeks and 6 months
Population: Data pertaining to 20 patients from each group were analysed after completing 6 months period
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | CAF+CTG+PRF | CAF+CTG
Number analyzed (Participants) | 20 | 20
mm
  Baseline | 4.5 [3 to 5.5] | 4 [3 to 5]
  6 weeks | 1 [1 to 3] | 2 [1 to 3]
  6 months | 1 [1 to 3] | 1.8 [1 to 3]
Statistical Analysis 1: Comparison: CAF+CTG+PRF vs CAF+CTG; Baseline; Test type: Superiority; p = 0.136, Mann-Whitney
Statistical Analysis 2: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 weeks; Test type: Superiority; p = 0.041, Mann-Whitney
Statistical Analysis 3: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 months; Test type: Superiority; p = 0.064, Mann-Whitney U — <0.05

5. Secondary Outcome: Keratinized Tissue Width
Description: measured from margin of the gingiva to mucogingival junction by periodontal probe
Time Frame: Baseline, 6 weeks and 6 months
Population: Data pertaining to 20 patients from each group were analysed after completing 6 months period
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | CAF+CTG+PRF | CAF+CTG
Number analyzed (Participants) | 20 | 20
mm
  Baseline | 3 [2 to 6] | 2.8 [2 to 6]
  6 weeks | 4 [2 to 7.5] | 3.5 [1.5 to 7]
  6 months | 4 [2 to 7.5] | 3.8 [2 to 7]
Statistical Analysis 1: Comparison: CAF+CTG+PRF vs CAF+CTG; Baseline; Test type: Superiority; p = 0.245, Mann-Whitney
Statistical Analysis 2: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 weeks; Test type: Superiority; p = 0.099, Mann-Whitney
Statistical Analysis 3: Comparison: CAF+CTG+PRF vs CAF+CTG; Test type: Superiority; p = 0.077, Mann-Whitney U

6. Secondary Outcome: Tissue Thickness
Description: under local anesthesia, measured from 1.5 mm below the margin of the gingiva with a spreader and its stopper silicon disc. Then, distance of the marked point was measured by using a standardized caliper to the closest 0.1 mm by periodontal probe
Time Frame: Baseline, 6 weeks and 6 months
Population: Data pertaining to 20 patients from each group were analysed after completing 6 months period
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | CAF+CTG+PRF | CAF+CTG
Number analyzed (Participants) | 20 | 20
mm
  Baseline | 0.9 [0.4 to 1.6] | 0.9 [0.4 to 1.6]
  6 weeks | 1.9 [1.4 to 2.6] | 1.6 [0.9 to 2.6]
  6 months | 1.9 [1.4 to 2.6] | 1.5 [1 to 2.2]
Statistical Analysis 1: Comparison: CAF+CTG+PRF vs CAF+CTG; Baseline; Test type: Superiority; p = 0.946, Mann-Whitney
Statistical Analysis 2: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 weeks; Test type: Superiority; p = 0.001, Mann-Whitney
Statistical Analysis 3: Comparison: CAF+CTG+PRF vs CAF+CTG; 6 months; Test type: Superiority; p = 0.001, Mann-Whitney U — <0.05

ADVERSE EVENTS:
Time Frame: 6 months
Description: At each visit, the patients were asked if they had such an experience of long-term swelling (more than 7 days), severe pain that did not response to analgesic consumption, ongoing bleeding (more than two days)
Arm/Group | PRF+CAF+CTG | CAF+CTG
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No